CLINICAL TRIAL: NCT05378867
Title: A Phase 3, Multicenter, Randomized and Double-blind Study Assessing the Interchangeability Between TRS003 and China-approved Bevacizumab® (Also Called China-approved Avastin) For First-Line Treatment of Patients With Metastatic Colorectal Cancer (CRC)
Brief Title: A Study Assessing the Interchangeability Between TRS003 and Bevacizumab® For CRC
Acronym: CRC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Teruisi Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRS00303002
Record Dates: First submitted 2022-04-21; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: A Phase 3, Multicenter, Randomized and Double-blind Study Assessing the Interchangeability between TRS003 and China-approved Bevacizumab® (also called China-approved Avastin) For First-Line Treatment of Patients with Metastatic Colorectal Cancer (CRC)
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study. Neither the subjects, nor the Investigator, nor the Sponsor knows which drug is being administered to which group. Only the Biostatistician who generated the actual randomization scheme with IWRS and the Pharmacist or nurse at the study center who prepares the study drugs and dose for the subjects will be unblinded. All other study related individuals including ancillary clinical staff, biological laboratory staff, clinical research associates, medical monitors, and scientific operation and management team at the study center will remain blinded to the treatment assignment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TRS003. (Experimental): Lead in Treatment Period
  * Will consist of 6 cycles of Bevacizumab® + mFOLFOX6
  * Each cycle length is 14 days
  After completion of the Lead-in Period, patients who have not progressed or experienced intolerable side effects and remain on study will be randomized 1:1 to either the Non-Switch or Switch Arm of the study.
  Switch Arm
  * TRS003, 5 mg/kg IV every 14 days with mFOLFOX6 for 1 cycle followed by switch to:
  * Bevacizumab®, 5 mg/kg IV every 14 days with mFOLFOX6 for 1 cycle followed by switch to:
  * TRS003, 5 mg/kg IV every 14 days with mFOLFOX6 until end of treatment due to PD, intolerability or other cause for stopping treatment. Intensive PK sampling will be performed after 7 cycles of this TRS003 switch period (to occur during Cycle 14, adequate for washout of preceding Bevacizumab®).
  Interventions: Biological: TRS003; Biological: China-approved Bevacizumab; Drug: mFOLFOX6
- China-approved Bevacizumab (Active Comparator): Lead in Treatment Period
  * Will consist of 6 cycles of Bevacizumab® + mFOLFOX6
  * Each cycle length is 14 days After completion of the Lead-in Period, patients who have not progressed or experienced intolerable side effects and remain on study will be randomized 1:1 to either the Non-Switch or Switch Arm of the study.
  Non-Switch Arm:
  * Bevacizumab®, 5 mg/kg administered IV every 14 days
  * mFOLFOX6 administered as described above every 14 days
  Interventions: Biological: China-approved Bevacizumab; Drug: mFOLFOX6

INTERVENTIONS:
Biological: TRS003 — * TRS003, 5 mg/kg IV every 14 days with mFOLFOX6 for 1 cycle followed by switch to:
  * Bevacizumab®, 5 mg/kg IV every 14 days with mFOLFOX6 for 1 cycle followed by switch to:
  * TRS003, 5 mg/kg IV every 14 days with mFOLFOX6 until end of treatment due to PD, intolerability or other cause for stopping treatment. Intensive PK sampling will be performed after 7 cycles of this TRS003 switch period
  Arms: TRS003.
Biological: China-approved Bevacizumab — • Bevacizumab®, 5 mg/kg IV every 14 days with mFOLFOX6 for 1 cycle
Drug: mFOLFOX6 — The mFOLFOX6 regimen is:
  * Oxaliplatin, 85 mg/m2 administered IV over 2 hours
  * LCV, 400 mg/m2 administered over 2 hours concurrent with oxaliplatin
  * 5-FU, 400 mg/m2 given as a slow IV push (bolus) over 5 minutes administered immediately after LCV
  * 5-FU, 2400 mg/m2 administered IV over 46 hours by infusion pump beginning immediately after FU IV bolus.

SUMMARY:
This is a Phase 3, multicenter, randomized and double-blind study assessing the interchangeability between TRS003 and China-approved Bevacizumab® (also called China-approved Avastin) for first-line treatment of patients with metastatic Colorectal Cancer (CRC), approximately 126 patients will be enrolled in this study. Patients who sign the informed consent, meet the eligibility criteria and are confirmed as non-progressors after lead-in treatment period with Bevacizumab® in combination with modified FOLFOX6 chemotherapy for 6 cycles, will be randomized (1:1) to either the non-switching arm and receive Bevacizumab® + modified FOLFOX6 for all subsequent cycles or to the switching arm and receive TRS003 alternating with Bevacizumab® in combination with mFOLFOX6 until disease progression or intolerability.

DETAILED DESCRIPTION:
This is a randomized, double-blind Phase 3 clinical trial evaluating the interchangeability, by a comparison of PK parameters between non-Switching and the Switching arms following the final switch between TRS003 and Bevacizumab® in patients with metastatic adenocarcinoma of the colon or rectum (please note that Bevacizumab® means China-approved Bevacizumab® in this protocol, unless otherwise specified). Approximately 126 patients will be enrolled in this study. Patients who sign the informed consent, meet the eligibility criteria and are confirmed as non-progressors after lead-in treatment period with Bevacizumab® in combination with modified FOLFOX6 chemotherapy for 6 cycles, will be randomized (1:1) to either the non-switching arm and receive Bevacizumab® + modified FOLFOX6 for all subsequent cycles or to the switching arm and receive TRS003 alternating with Bevacizumab® in combination with mFOLFOX6 until disease progression or intolerability. There will be 3 switches as detailed in the Treatment section (below) and the Schema. If oxaliplatin-induced neurotoxicity requires discontinuation of oxaliplatin, treatment will continue using leucovorin (LCV) plus 5-fluorouracil (5-FU) in combination with either Bevacizumab® or TRS003 until progressive disease (PD), intolerability, or other cause for stopping treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented adenocarcinoma of the colon or rectum
2. Must have radiographic documentation of measurable metastatic disease (per RECIST v1.1)
3. Patients with resected primary tumors are eligible if documented metastatic disease is present.
4. Age ≥ 18 years
5. ECOG Performance Status of 0-1
6. Patients who received oxaliplatin/fluorouracil-based adjuvant chemotherapy then developed metastatic disease are eligible if > 12 months since last adjuvant chemotherapy treatment. Consider biopsy to confirm lesions are metastatic colorectal cancer, especially if initial CRC was stage I.
7. May have received radiation with radio-sensitizing chemotherapy if completed > 12 months before enrollment. Patients with rectal cancer who have received locoregional radiation therapy are eligible if they have measurable metastatic disease that is outside the radiation therapy portal.
8. Patients with left or right sided primary colon cancers are eligible as are patients with RAS or BRAF mutant tumor (molecular determination is not required).
9. Hypertension must be well controlled (< 150/90) on a stable anti-hypertensive regimen.
10. Patients on full-dose anticoagulation or taking anti-platelet agents are eligible if on a stable dose of medication and have no active bleeding or conditions that predispose to bleeding.
11. For women of childbearing potential, must consent to use two highly effective methods (i.e., total abstinence, placement of an intrauterine device) of contraception during treatment and for an additional 90 days after the last administration of study drug.

    Men with a partner of childbearing potential, must consent to use two highly effective methods of contraception during treatment and for an additional 90 days after the last administration of study drug.
12. Required laboratory values:

    * Granulocytes ≥ 1500/uL
    * Hemoglobin ≥ 9.0 grams/dL
    * Platelets ≥ 100,000/uL
    * Serum creatinine < 1.5 × ULN or calculated creatinine clearance (CLcr) > 50 mL/min.
    * Total bilirubin ≤ 1.5 × upper limit of normal (ULN) except for patients with Gilbert's syndrome, who are included if total bilirubin is < 3 × ULN or if direct bilirubin is < 1.5 × ULN.
    * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 × ULN. For those with hepatic metastases, AST and ALT ≤ 5 × ULN.
    * Albumin ≥ 2.5 g/dL
    * Urinalysis ≤ 1+ protein. Patients that have ≥ 2+ proteinuria must have < 1g of protein on a 24h urine collection.

Exclusion Criteria:

1. Prior systemic or regional treatment for metastatic disease
2. Prior exposure to drugs that target VEGF or VEGF receptors (e.g., tyrosine kinase inhibitors, monoclonal antibodies, or soluble receptors).
3. Patients whose tumors have microsatellite instability-high or mismatch repair deficiency
4. Radiotherapy to greater than 25% of the bone marrow. Standard adjuvant rectal cancer chemoradiation will not exclude the patient.
5. Previous or concurrent malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer that the patient has been disease-free for 5 years
6. Sensory or peripheral neuropathy of ≥ grade 2 at baseline
7. Known central nervous system metastases or carcinomatous meningitis
8. Interstitial pneumonia or medically significant interstitial fibrosis of the lung
9. Pleural effusion or ascites that causes ≥ grade 2 dyspnea.
10. Colon or small bowel disorders with baseline symptoms including 3 watery or soft stools per day (patients without colostomy or ileostomy; patients with stoma may be entered at Investigator's discretion).
11. Uncontrolled seizure disorder or active neurological disease
12. Current congestive heart failure (NY Heart Association Class II, III, or IV)
13. Significant hemorrhagic events within 6 months prior to the study screening including hemoptysis > 2.5 mL of red blood, gastrointestinal bleeding, hematemesis, central nervous system hemorrhage, severe epistaxis or vaginal bleeding, etc.
14. Venous or arterial thrombotic events within 6 months of enrollment, including pulmonary embolism or deep vein thrombosis, transient ischemic attack (TIA), cerebrovascular accident (CVA), unstable angina, or myocardial infarction (MI) requiring surgical or medical intervention. Patients with clinically significant peripheral vascular disease or any other arterial thrombotic event are ineligible.
15. Serious or non-healing wound, ulcer, or bone fracture.
16. Any major surgical procedure within 28 days prior to screening or anticipated elective surgery during the study. Any minor surgery such as central vein catheterization within 48 hours prior to the first dose of the study drugs.
17. Hypersensitivity to Chinese hamster ovary cell products or to recombinant human or murine antibodies.
18. Hypersensitivity to oxaliplatin or any other platinum-based drug.
19. Active hepatitis B or hepatitis C virus. Patients with evidence of infection with hepatitis B who have an undetectable viral load are eligible for study entry. Patients with evidence of infection with hepatitis C should have completed curative therapy.
20. History of HIV infection.
21. Pregnant or breast-feeding females
22. Any uncontrolled intercurrent illness or condition that in the judgement of the Investigator may endanger the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
AUCtau，Area under the curve over the dosing interval | Cycle 14 (each cycle is 14 days)
  The natural log-transformed AUCtau in Cycle 14 will be analyzed.

SECONDARY OUTCOMES:
C trough， trough concentration | Cycle 14 (each cycle is 14 days)
  Besides AUCtau, the PK parameters to be estimated will include the trough concentration (Ctrough), the maximum concentration (Cmax), and time to reach Cmax (Tmax).
C max，maximum concentration | Cycle 14 (each cycle is 14 days)
  Besides AUCtau, the PK parameters to be estimated will include the trough concentration (Ctrough), the maximum concentration (Cmax), and time to reach Cmax (Tmax).
T max，the time to reach Cmax | Cycle 14 (each cycle is 14 days)
  Besides AUCtau, the PK parameters to be estimated will include the trough concentration (Ctrough), the maximum concentration (Cmax), and time to reach Cmax (Tmax).
ADA，anti-drug antibody | at Day 1 of every 2 cycles（each cycle is 14 days）
  anti-drug antibody (ADA) and neutralizing antibody if ADA is positive
PFS，Progression-free survival | Cycle 14 (each cycle is 14 days)
  Progression-free survival (PFS) is defined as the time from randomization to Investigator-determined PD or death due to any cause in the absence of documented PD.
OS，Overall survival | Cycle 14 (each cycle is 14 days)
  Overall survival (OS) is defined as the time from randomization to death due to any cause.
ORR，objective response rate | Cycle 14 (each cycle is 14 days)
  ORR in the TRS003 Arm/ORR in the China-approved bevacizumab Arm Confidence interval of ORR in each group will be estimated by the Clopper-Pearson Exact method.
DOR，Duration of response | Cycle 14 (each cycle is 14 days)
  Duration of response (DOR) is defined as the time from the date of the first documentation of Investigator-determined response in patients with confirmed objective tumor response (CR or PR) to the first documentation of Investigator determined disease progression (PD) or to death due to any cause in the absence of documented PD.

IPD SHARING:
Plan to Share IPD: No